CLINICAL TRIAL: NCT07164300
Title: Comparative Study of Tranexamic Acid Dosage Regimens in Patients Undergoing Cardiac Surgery Under Cardiopulmonary Bypass
Brief Title: Comparative Study of Tranexamic Acid Dosing in Cardiac Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Evangelia Samara, Assistant Professor of Anaesthesiology, University of Ioannina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 886/11-11-2024
Record Dates: First submitted 2025-08-07; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Blood Coagulation Disorder; Postoperative Blood Loss; Adverse Drug Event; Fibrinolysis; Hemorrhage; Tranexamic Acid Adverse Reaction
MeSH Terms: conditions — Blood Coagulation Disorders; Postoperative Hemorrhage; Drug-Related Side Effects and Adverse Reactions; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Group 1 will receive a tranexamic acid dosage of 10mg/kg prior to operation start, followed by transfusion rate of 1mg/kg/h until the end of the surgery.
  Interventions: Drug: Tranexamic acid at a dose of 10 mg/kg followed by 1 mg/kg/h
- Group 2 (Experimental): Group 2 will receive a tranexamic acid dosage of 20mg/kg prior to operation start.
  Interventions: Drug: Tranexamic acid at a dose of 20 mg/kg
- Group 3 (Experimental): Group 3 will receive a tranexamic acid dosage of 30mg/kg prior to operation start.
  Interventions: Drug: Tranexamic acid at a dose of 30 mg/kg

INTERVENTIONS:
Drug: Tranexamic acid at a dose of 10 mg/kg followed by 1 mg/kg/h — Group 1: administration of tranexamic acid at a dose of 10 mg/kg followed by 1 mg/kg/h
  Other Names: Group 1
  Arms: Group 1
Drug: Tranexamic acid at a dose of 20 mg/kg — Group 2: administration of tranexamic acid at a dose of 20 mg/kg
  Other Names: Group 2
  Arms: Group 2
Drug: Tranexamic acid at a dose of 30 mg/kg — Group 3: administration of tranexamic acid at a dose of 30 mg/kg
  Other Names: Group 3
  Arms: Group 3

SUMMARY:
Tranexamic axid is routinely used as an antifibrinolytic agent in cardiac surgery to reduce the risk of blood loss and transfusion. However, there is no consensus regarding the dosage regimen of tranexamic acid that should be administered. The purpose of this study is to compare different dosages of tranexamic acid in cardiac surgery using cardiopulmonary bypass regarding the duration of inhibition of fibrinolysis as measured by the ClotPro test.

Blood samples will be taken from the arterial line placed in the patient at specified time points in order to perform viscoelastic tests (ClotPro, TPA test), to detect successful inhibition of fibrinolysis and to measure tranexamic acid levels in the patient's blood. In case the action of tranexamic acid stops early postoperatively an additional dose of the medication will be administered to the patient.

DETAILED DESCRIPTION:
Excessive bleeding and blood transfusions are common in patients undergoing cardiac surgery. Antifibrinolytic therapy reduces the risk of blood loss and transfusion among patients undergoing cardiac surgery. Tranexamic acid is an antifibrinolytic agent that forms a reversible complex with plasminogen. Guidelines for the management of bleeding in patients recommend the routine use of tranexamic acid for cardiac surgery in adults. However, there is no consensus regarding the dosage regimen of tranexamic acid that should be administered. More specifically, several dosage regimens have been studied in the literature. Although higher doses of tranexamic acid achieve a marginal reduction in postoperative bleeding, they increase the risk of drug-related postoperative complications. Based on a recent 2021 meta -analysis, it appears that lower doses of tranexamic acid (eg 20 mg / kg or 10mg/kg followed by 1mg kg-1 h-1) are safe and effective. In the literature, the duration of inhibition of fibrinolysis after the administration of tranexamic acid has been studied using the point of care test ClotPro (a thromboelastometry analyzer) in relatively large dosages (total dose: 50 mg / kg), while there are no relevant randomized clinical studies. Lower doses of tranexamic acid have been shown to be effective and safe, although their duration of action has not been studied using the viscoelastic Clot Pro-TPA test and their correlation with blood tranexamic acid concentration.

The present study aims to evaluate different dosages of tranexamic acid in cardiac surgery using cardiopulmonary bypass. The primary outcome is the duration of inhibition of fibrinolysis as measured by the ClotPro test and the correlation of imprinting with tranexamic blood concentration.

Methods:

Perioperative management will follow standard department practice. Patients for elective cardiac surgery using cardiopulmonary bypass will be randomized to receive tranexamic acid after induction of anesthesia at three different doses of 30 mg / kg , 20 mg / kg or 10 mg / kg followed by 1 mg / kg / h until the end of the surgery. All patients will sign an informed consent prior to their inclusion in the study.

Data collection:

During pre-operative evaluation, age, weight, height, sex, BSA, ASA classification, Euroscore II, standard perioperative laboratory testing results, medication and co-morbidities will be documented.

Intraoperatively, the duration of anesthesia, the type and duration of surgery, the cardiopulmonary bypass and aortic cross clamping time will be documented, as well as drugs administered and related adverse events.

At specified time points (during induction of anesthesia and before administration of the drug, after the completion of the single administration, after the end of the cardiopulmonary bypass, six and twelve hours after the administration of the drug and then twelve hours until the values ML and LT in the TPA test to be greater than 50% and less than 2100 sec respectively) blood samples will be taken from the arterial line placed in the patient. The purpose will be to perform viscoelastic tests (ClotPro , TPA test), to detect successful fibrinolysis inhibition and measure tranexamic acid levels in the patient's blood. In case the ML and LT values are as above before or at the six-hour sample, the patient will be given an additional 10 mg/kg and the measurements will be repeated.

Also, the total administration of blood and products, the administration of coagulation factors intraoperatively and during the ICU stay, as well as the total postoperative bleeding in the first 24 hours are recorded. The need for reoperation due to postoperative bleeding, seizures, and all serious adverse events related to surgery and general anesthesian and/or the tranexamic acid administration in the postoperative period are also recorded.

Postoperatively, the duration of mechanical ventilation and sedation in the Cardiac Surgery ICU, the length of stay in the Cardiac Surgery ICU, the length of stay in the Hospital before surgery and after discharge from the Cardiac Surgery ICU, and all - cause in hospital mortality will be recorded.

The present study aims to evaluate different dosages of tranexamic acid in cardiac surgery using cardiopulmonary bypass. It is a prospective, randomized, comparative study. The primary outcome is the duration of inhibition of fibrinolysis as measured by the ClotPro test and the correlation of imprinting with tranexamic blood concentration. Secondary outcomes are blood and blood product transfusion, need of coagulation factors administration, postoperative bleeding, time of mechanical ventilation, length of stay in the Intensive Care Unit (ICU), total length of hospitalization and all - cause in hospital mortality. Also, secondary outcomes include the correlation of tranexamic acid dosage with the postoperative incidence of seizures and thrombotic complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective cardiac surgery using cardiopulmonary bypass
* Patients to have discontinued anticoagulant and antiplatelet therapy preoperatively according to guidelines.

Exclusion Criteria:

* Age below 18 years
* Patient refusal
* Pregnancy
* End-stage renal disease
* History of epilepsy,
* Cardiac surgery without the use of cardiopulmonary bypass (off-pump)
* Emergency operations
* Known allergy to the administered agents.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
duration of inhibition of fibrinolysis as measured by the ClotPro-TPA test | time(hours) from tranexamic acid administration until the values of ML and LT in the TPA test (Clot Pro) become greater than 50% and less than 2100 sec, respectively,up to 240 hours post tranexamic acid bolus administration.
  time(hours) from tranexamic acid administration until the values of ML and LT in the TPA test (Clot Pro) become greater than 50% and less than 2100 sec, respectively (0,3,6,12,24,36,48 etc up to 240 hours post tranexamic acid bolus administration).
tranexamic blood concentration | time(hours) from tranexamic acid administration until the values of ML and LT in the TPA test (Clot Pro) become greater than 50% and less than 2100 sec, respectively, and up to up to 240 hours post tranexamic acid bolus administration.
  Blood concentration of tranexamic acid at predifined study time points (0,3,6,12,24,36,48 etc up to 240 hours post tranexamic acid bolus administration)

SECONDARY OUTCOMES:
transfusion of blood and products | Ιntraoperatively and during the first 24 hours postoperatively
  Patient's transfusion requirements for packed red blood cell units, fresh frozen plasma units and platelets units.
need of administration of coagulation factors | intraoperatively and during the first 24 hours postoperatively
  Need for administration of coagulation factors such as fibrinogen (gr), prothrombin complex concentrate, PCC (IU) and calcium (gr)
Postoperative bleeding | During the first 24 hours postoperatively
  The total amount of blood present in the drainage tube in ml.
reoperation | From the end of surgery until the patient's discharge from the hospital or death (up to 1 year)
  The need for reoperation due to postoperative bleeding
Mechanical ventilation | From the end of surgery until the patient's extubation, or patient's death if not extubated. (up to 1 year)
  The duration of postoperative mechanical ventilation in hours.
Length of stay in the Intensive Care Unit | From the end of surgery until the patient's discharge from the ICU, or patient's death if not discharged. (up to 1 year)
  The duration of the patient's stay in the ICU in hours.
Length of hospitalization | From the day of surgery until the patient's discharge from the hospital, or patient's death if not discharged. (up to 1 year)
  The total duration of the patient's hospital stay in days
All cause in-hospital mortality | From the day of surgery until the patient's discharge from the hospital (up to 1 year)
  All causes of the patient's death during their hospital stay are recorded.
postoperative incidence of seizures | From the administration of tranexamic acid until the patient's discharge from the hospital (up to 1 month)
  The correlation between the dosage of tranexamic acid and the postoperative incidence of seizures.
thrombotic episodes | From the administration of tranexamic acid until the patient's discharge from the hospital. (up to one month)
  The correlation between the dosage of tranexamic acid and the postoperative incidence of thrombotic events.

CONTACTS AND LOCATIONS:
Overall Officials: Evangelia Samara, Principal Investigator — University of Ioannina
Locations (1):
- University Hospital of Ioannina, Ioannina, Greece

IPD SHARING:
Plan to Share IPD: No